CLINICAL TRIAL: NCT06333912
Title: Accuracy of Novel Ridge Splitting Guide Design in Comparison to Freehand With Simultaneous Implant Placement
Brief Title: Accuracy of Guided Ridge Splitting With Simultaneous Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ridgesplittingguided
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Dental Implant
Keywords: guided ridge splitting, atrophic maxilla, osseodensification drills.
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group treated with guided ridge splitting. (Experimental): virtual surgical planning using planning software Blue Sky Bio (BSB) and 3D printed surgical guide are fabricated to guide the ridge splitting procedure and implant drilling and placement.
  Interventions: Procedure: dental implant placement with ridge splitting.
- control group treated with conventional ridge splitting. (Active Comparator): Freehand surgery is done including ridge splitting and implant plaement
  Interventions: Procedure: dental implant placement with ridge splitting.

INTERVENTIONS:
Procedure: dental implant placement with ridge splitting. — ridge splitting to increase bone width in atrophic maxilla with simultaneous implant placement

SUMMARY:
Assessing whether is there a difference between computer-guided ridge splitting and conventional technique with simultaneous implant placement in patients with maxillary width deficiency.

DETAILED DESCRIPTION:
Two groups one treated with ridge splitting using guided surgery and the other one treated with freehand surgery and both groups had simultaneous dental implants the first one had guided placement and the other one was freehand.

ELIGIBILITY:
Inclusion Criteria:

* Patient with missing maxillary anteriors or premolars teeth.
* Tooth extraction at the implant sites was performed at least 4 months before the surgery.
* The bone width of the crestal one -third (3-5 mm) with sufficient bone height allowing for simultaneous implant placement.
* Free from any systemic disease or local pathological lesions that may affect bone healing or contraindicate implant placement.
* With no history of any previous grafting surgeries at the area of interest.

Exclusion Criteria:

* Sever concavity of the alveolar ridge.
* Bad oral hygiene ( Silness-Löe index (score 2-3).
* Heavy smoker (smoke greater than or equal 25 cigarettes per day).
* Presence of acute infections or periapical lesions in adjacent teeth.
* Parafunctional habits.
* Pregnant females.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Assessing the accuracy of guided surgery | one week
  superimposition of post-op cbct to the planned position to check the accuracy of implant positions.

SECONDARY OUTCOMES:
the bone-width increase between control and study group. | 6 months
  evaluation of two techniques of ridge splitting in increasing bone width.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elbayaa, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Faculty of dentistry, Alexandria, Egypt